CLINICAL TRIAL: NCT04096833
Title: The Effect of Virtual Reality Versus Standard-of-care Treatment on Pain Perception During Paediatric Vaccination: Study Protocol for a Randomised Controlled Trial.
Brief Title: Virtual Reality for the Treatment of Pain in Pediatric Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Laura García Garcés, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CardenalHU_Nursing
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Virtual Reality; Vaccination; Pain; Nursing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the care giver (nurse) will know the assignment of participants to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants use as a distracting measure Virtual Reality glasses during the vaccination.
  Interventions: Other: Virtual Reality Group
- Control Group (No Intervention): Participants use usual non-virtual distracting measures during the vaccination.

INTERVENTIONS:
Other: Virtual Reality Group — Participants are from 3 to 14 years old who attend a pediatric primarey health care of the Fuensanta Health Center (Valencia) for immunization by vaccine.
  Arms: Intervention Group

SUMMARY:
Objective: to estimate the effect of virtual reality as a distracting technique against traditional distracting techniques in the vaccination procedure in the pediatric population.

Design: randomized clinical trial. Field of study: the study will be carried out in the field of pediatric primary care nursing consultation, where the pediatric systematic vaccination is performed.

Subjects to study: the sample will be made up of children from 3 to 14 years old who are punctured for immunization in the Fuensanta Health Center that belongs to the Department of Health Valencia-General Hospital.

Variables: age, sex, family country of origin, years living in Spain, number of children of the nuclear family, order in the number of siblings, socioeconomic level, age of the caregiver that accompanies the child, affiliation / bond with the child . Group to which the subject belongs (intervention group vs. control group). Number of punctures received in the last year. Heart rate pre and post vaccination. Type of vaccine. Combination of several punctures in the query. Previous use of virtual reality. Level of pain and fear after puncture. Parent or legal guardian satisfaction.

Data collection: it will be held at the Health Center on the same day as the vaccination prodecure. On the part of the nurse (heart rate, type of vaccine, combination of several punctures), the child (pain, fear) and the parents / legal guardian (satisfaction, sociodemographic).

Data analysis: The descriptive analysis of the quantitative variables will be carried out through the calculation of means, typical deviations, medians, ranges, minimum and maximum values. Qualitative variables will be analyzed in absolute and relative frequencies. For the statistical inference analysis, the T-test analysis of mean difference or U-Mann Whitney (according to normal compliance) will be used. All analyzes will be performed with a 95% confidence interval.

DETAILED DESCRIPTION:
Process:

The health professional responsible for carrying out the intervention will be the nurse of the pediatric consultation of the Health Center where the study will be carried out. She is the only nurse in this center, so she will be the only professional to perform the procedure on all subjects participating in the study; in this way the variability in the puncture technique is avoided.

The nurse will recruit potential participants who meet inclusion criteria, informing about the research and answering their possible questions. Once participants wishing to be part of the study have signed the informed consent, they will be coded by numbers. These numerical codes will be linked chronologically to the random sequence previously generated by the sealedenvelopeTM software. Once the nurse knows the group to which the participant belongs, she will perform the corresponding intervention.

The evaluation after the completion of the vaccination procedure will be carried out through self-administered scales (by the child for pain and fear variables, and by the caregiver for sociodemographic and satisfaction variables). In addition, the nurse will record data regarding vaccinations.

The data collection time is estimated at 1 year and a half or until the sample size is reached.

Intervention:

The study groups will be determined by the randomization of the sample into two groups: GI and GC. The GI will use as a distracting measure the viewing of VR experiences adapted to their age with the Oculus Go VR glasses during the puncture. The GC will use habitual non-virtual distracting measures: being in the arms of the main caregiver or maintaining physical contact with him (for example, shaking hands) and / or playing or watching videos with the mobile phone of the parents or legal guardian.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 and 14 years old, who attend a pediatric nursing office of the Fuensanta Health Center (Valencia) for immunization by vaccine.
* Children who are accompanied by a caregiver (father, mother, legal guardian) during the procedure.
* That both the child and the caregiver understand and speak Spanish.
* That they have consented to participate in the study: in children by verbal consent and in their father, mother, legal guardian, by signing the informed consent document.

Exclusion Criteria:

* Children with sensory problems that prevent the use of RV.
* Children with sensory impairment of pain perception (for example, spina bifida).
* Children who have taken analgesic medication on the day of the puncture, either orally or topically in the puncture area.
* Children with a history of seizures or dizziness.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Compare the perception of pain in children during the vaccination between participants to recive virtual reality and to recive usual distraction mesures: Wong-Baker FACES scale | It is immediately after vaccination.
  El dolor es una experiencia emocional y sensorial desagradable, que puede deberse a un procedimiento terapéutico como la vacunación. Para medir el nivel de dolor del niño después de la vacunación, se utilizará la Escala de calificación del dolor: escala FACES de Wong-Baker. Es un cuestionario validado desarrollado por Bieri en 1990. Está indicado para niños entre 3 y 18 años. La escala va de 0 a 10 y tiene 6 caras. A cada cara se le asigna un puntaje. El primero, con un valor de 0, equivale a "no hurt"; la segunda, con un valor de 2 , equivale a "hurts little bit", el tercero, con un valor de 4 es igual a "hurts little more", el cuarto, con un valor de 6, significa "hurts even more", el quinto, con un valor de 8, es igual a "hurts whole lot" y el último, con un valor de 10 es igual a "hurts worse". Se le pide al paciente que seleccione la cara que mejor describa cómo se siente. En el nivel psicométrico, esta escala se valida r = .90, alfa de Cronbach = .93 (Keck, 1996).

SECONDARY OUTCOMES:
Compare the perception of fear in children during the vaccination between participants to recive virtual reality and usual distraction mesures. | It is immediately after vaccination.
  Vaccination causes fear in children. To assess the fear perceived by the child, the Child Fear Scale (CFS) will be used (McMurtry, Noel, Chambers, McGrath, 2011). CFS consists of five faces that show different levels of fear: the first face, no. 0, the second, no. 1, the third, no. 2, the fourth, no. 3, and the last, no. 4. The first face equals "no fear" and the last "maximum fear possible". The CFS is an effective instrument for measuring fear related to pain during vaccination of children. This tool is validated (Interrater Time 1 reliability: rs = .51, p <.001 and test-retest reliability rs = .76, p <.001).

OTHER OUTCOMES:
Compare the satisfaction of caregiver (mothers, fathers and legal guardians) satisfaction during the vaccination between participants: questionnaire | It is immediately after vaccination.
  Caregivers (mothers, fathers and legal guardians) will complete a satisfaction questionnaire prepared by Gold and Mahrer (2018) to assess satisfaction with the vaccination procedure and with the distraction measures used (RV or habitual distraction measures). This questionnaire has 11 items, 9 of them with a Likert scale ranging from 1 to 10. 1 equals "not at all", "not at all well" or "nothing more". 5 equals "somewhat", moderately well "," moderatly "or" some things more. "10 equals" definitely "," extremely well "," extremely "or" a lot more. "The first and last question of the questionnaire are open questions and the sixth question is a docotomic answer: yes / no This tool is not validated.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad CEU-Cardenal Herrera, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Keck JF, Gerkensmeyer JE, Joyce BA, Schade JG. Reliability and validity of the Faces and Word Descriptor Scales to measure procedural pain. J Pediatr Nurs. 1996 Dec;11(6):368-74. doi: 10.1016/S0882-5963(96)80081-9. PMID 8991337
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848